CLINICAL TRIAL: NCT00796302
Title: Stimulant and Risperidone in Children With Severe Physical Aggression
Brief Title: Treatment of Severe Childhood Aggression (The TOSCA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Aman (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Michael Aman, Retiree-Faculty, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH077907 (NIH); DSIR 84-CTS; 1R01MH077907-01A2 (NIH); 1R01MH077676-01A2 (NIH); 1R01MH077750-01A2 (NIH); 1R01MH077997-01A2 (NIH)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Conduct Disorder; Attention Deficit and Disruptive Behavior Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Conduct Disorder; Attention Deficit and Disruptive Behavior Disorders | interventions — Methylphenidate; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Children will receive active methylphenidate HCl and active risperidone. Parents will receive parent management training.
  Interventions: Drug: Methylphenidate HCl; Drug: Risperidone; Behavioral: Parent Management Training (PMT)
- 2 (Active Comparator): Children will receive methylphenidate HCl and placebo instead of the active risperidone. Parents will receive parent management training.
  Interventions: Drug: Methylphenidate HCl; Behavioral: Parent Management Training (PMT); Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate HCl — For children weighing less than 25 kg, the dose will be titrated at 18 mg for the first 7 days, 36 mg for the next 4 days, and, if needed, 54 mg for the next 4 days. For children weighing more than 25 kg, the dose will be titrated at 18 mg for the first 4 days, 36 mg for the next 3 days, 54 mg for the next 4 days, and 72 mg for the next 3 days.
  Once the child's optimal dose is established, he or she will continue on that dose for the rest of the 21-week trial.
  One pill is taken once daily.
  Other Names: Concerta
Drug: Risperidone — For children weighing less than 45 kg, the dose will start at 0.5 mg at night. After 4 days, the child's dose may be increased to 1 mg a day. On Day 8, the child's dose may be increased to 1.5 mg a day. On Day 16, the child's dose may be increased to 2.0 mg a day. On Day 22, the child's dose may be increased to 2.5 mg a day.
  For children weighing more than 45 kg, the dose will start at 0.5 mg at night. After 4 days, the child's dose may be increased to 1.0 mg a day. On Day 8, the child's dose may be increased to 1.5 mg a day. On Day 12, the child's dose may be increased to 2.0 mg a day. On Day 15, the child's dose may be increased to 2.5 mg a day. On Day 18, the child's dose may be increased to 3 mg a day. On Day 23, the child's dose may be increased to 3.5 mg a day.
  Other Names: Risperdal
  Arms: 1
Behavioral: Parent Management Training (PMT) — PMT will include individual parent sessions held weekly for 9 weeks, with two booster sessions to be completed during the 3-month extension. Sessions will include development of problem-solving skills and behavior management strategies, practice activities, and role-playing with the behavioral therapist.
  Other Names: Community Parent Education Program
Drug: Placebo — One pill will be taken once daily for the first 4 days and then twice daily until Week 21.
  Arms: 2

SUMMARY:
This study will determine the safety and effectiveness of two medications for treating aggression in children with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
ADHD is characterized by inattention, impulsivity, and hyperactivity. Children with ADHD sometimes also have disruptive behavior disorders (DBDs), such as conduct disorder (CD), which is estimated to develop in 20% to 40% of children with ADHD, and oppositional defiant disorder (ODD), which is estimated to develop in 33% to 50% of children with ADHD. These two disorders place youth at risk of other psychiatric disorders, especially substance abuse disorders. Several medications have been tested to treat conduct disorders in aggressive children, and, among these, risperidone and methylphenidate hydrochloride (HCl) have relatively good records of safety and tolerability. Psychostimulants, such as methylphenidate HCl, can reduce the symptoms in some, but not all, children with DBDs. Combining methylphenidate HCl with risperidone may be one way to increase the effectiveness of drug treatments. This study will compare the effectiveness of methylphenidate HCl alone versus methylphenidate HCl combined with risperidone for treating aggressive behavior in children with ADHD. Participation in this study will last 1 year. The child participant and a parent will attend all study visits. Two initial visits will involve a battery of baseline tests, including a psychological clinical interview, physical examination, lab tests, and an electrocardiogram (ECG). The parents will undergo a parent education session and complete questionnaires about their child's behavior, emotions, and medication side effects. The child will have his or her vital signs measured and complete tests of verbal memory and attention and impulsiveness. After the second visit, the child participant will be randomly assigned to receive either methylphenidate HCl alone or methylphenidate HCl plus risperidone.

For the next 3 weeks, all child participants will take methylphenidate HCl at a dose that will start low and gradually be increased until the most effective dose is determined. For the next 6 weeks, child participants will add either risperidone or a placebo to their regimen of methylphenidate HCl. This second medication will also be started at a low dose and raised to appropriate levels of tolerability. During the 9 weeks of medication adjustment, participants will attend weekly study visits to complete questionnaires and have their vital signs measured. Parents will attend education sessions at each of these visits. The child's teacher will also fill out weekly questionnaires on the child's behavior. Every 3 weeks, child participants will be tested on verbal memory, attention, and impulsiveness. After the 9-week period, child participants will again undergo a physical exam, lab tests, and an ECG.

At this point, if the child's behavior has improved, the child will continue the same treatment for the next 3 months. Monthly study visits will include parent education sessions and recording of parent and teacher evaluations of the child. All participants will attend a 1-year follow-up visit that will include previous assessments.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of ADHD, any subtype
* DSM-IV diagnosis of a disruptive behavior disorder, including CD or ODD
* Evidence of serious physical aggression, as rated on the Overt Aggression Scale-Modified, and as determined by parent or guardian ratings on the NCBRF D-Total Score. In addition, the blinded clinician must assign a clinical global impressions severity score of 4 or greater for aggression.
* Prior to random assignment, participants must be free of all psychotropic medicines for 2 weeks for most drugs (such as most antidepressants, alpha agonists, beta blockers, anxiolytics, mood stabilizers, and antihistamines), and 4 weeks for depot antipsychotics and fluoxetine.

Exclusion Criteria:

* Full-scale IQ below 71
* Pregnancy or a history of seizure disorder or other neurological or medical disorders for which medication may present a considerable risk
* Abnormal liver function
* Pervasive developmental disorder, schizophrenia or other psychotic disorders, or eating disorders
* Currently taking other psychotropic medications from which discontinuation would present a significant risk. Participants may not discontinue a satisfactory medication to participate.
* Presence or history of major depressive disorder
* Diagnosis of bipolar disorder
* A hypomanic/biphasic score of 36 or greater as rated by child's parent on the General Behavior Inventory and confirmed by clinician as indication of mood disorder
* Active substance abuse disorder or lack of control of substance use that does not allow for safe medication administration
* Evidence of current child abuse or neglect
* History of suicide attempt in the past year or current suicidal ideation with plan and/or intent
* Family history of type II diabetes in two or more first degree relatives, defined as biological parents and/or full biological siblings

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2008-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Aman, PhD, Principal Investigator — Ohio State University; Oscar G. Bukstein, MD, MPH, Principal Investigator — University of Pittsburgh; Kenneth D. Gadow, PhD, Principal Investigator — State University of New York Stony Brook; Robert L. Findling, MD, Principal Investigator — Case Western Reserve University
Locations (4):
- United States (4):
  - State University of New York Stony Brook, Stony Brook, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Nisonger Center, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Aman MG, Bukstein OG, Gadow KD, Arnold LE, Molina BS, McNamara NK, Rundberg-Rivera EV, Li X, Kipp H, Schneider J, Butter EM, Baker J, Sprafkin J, Rice RR Jr, Bangalore SS, Farmer CA, Austin AB, Buchan-Page KA, Brown NV, Hurt EA, Grondhuis SN, Findling RL. What does risperidone add to parent training and stimulant for severe aggression in child attention-deficit/hyperactivity disorder? J Am Acad Child Adolesc Psychiatry. 2014 Jan;53(1):47-60.e1. doi: 10.1016/j.jaac.2013.09.022. Epub 2013 Nov 18. PMID 24342385
- [Result] Kaat A, Farmer C, Gadow K, Findling RL, Bukstein O, Arnold LE, Bangalore S, McNamara N, Aman M. Factor Validity of a Proactive and Reactive Aggression Rating Scale. J Child Fam Stud. 2015 Sep 1;24(9):2734-2744. doi: 10.1007/s10826-014-0075-5. Epub 2014 Nov 27. PMID 26504369
- [Result] Farmer CA, Brown NV, Gadow KD, Arnold LE, Kolko DG, Findling RL, Molina BS, Buchan-Page KA, Rice RR Jr, Bangalore SS, Bukstein O, Rundberg-Rivera EV, McNamara N, Aman MG. Comorbid symptomatology moderates response to risperidone, stimulant, and parent training in children with severe aggression, disruptive behavior disorder, and attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2015 Apr;25(3):213-24. doi: 10.1089/cap.2014.0109. PMID 25885011
- [Result] Rundberg-Rivera EV, Townsend LD, Schneider J, Farmer CA, Molina BB, Findling RL, Gadow KD, Bukstein OG, Arnold LE, Kolko DJ, Buchan-Page KA, McNamara NK, Michel C, Austin A, Kipp H, Rice RR, Aman MG. Participant satisfaction in a study of stimulant, parent training, and risperidone in children with severe physical aggression. J Child Adolesc Psychopharmacol. 2015 Apr;25(3):225-33. doi: 10.1089/cap.2014.0097. PMID 25885012
- [Result] Arnold LE, Gadow KD, Farmer CA, Findling RL, Bukstein O, Molina BS, Brown NV, Li X, Rundberg-Rivera EV, Bangalore S, Buchan-Page K, Hurt EA, Rice R, McNamara NK, Aman MG. Comorbid anxiety and social avoidance in treatment of severe childhood aggression: response to adding risperidone to stimulant and parent training; mediation of disruptive symptom response. J Child Adolesc Psychopharmacol. 2015 Apr;25(3):203-12. doi: 10.1089/cap.2014.0104. PMID 25885010
- [Result] Gadow KD, Arnold LE, Molina BS, Findling RL, Bukstein OG, Brown NV, McNamara NK, Rundberg-Rivera EV, Li X, Kipp HL, Schneider J, Farmer CA, Baker JL, Sprafkin J, Rice RR Jr, Bangalore SS, Butter EM, Buchan-Page KA, Hurt EA, Austin AB, Grondhuis SN, Aman MG. Risperidone added to parent training and stimulant medication: effects on attention-deficit/hyperactivity disorder, oppositional defiant disorder, conduct disorder, and peer aggression. J Am Acad Child Adolesc Psychiatry. 2014 Sep;53(9):948-959.e1. doi: 10.1016/j.jaac.2014.05.008. Epub 2014 Jun 12. PMID 25151418
- [Derived] Grondhuis SN, Farmer CA, Arnold LE, Gadow KD, Findling RL, Molina BSG, Kolko DJ, Buchan-Page KA, Rice RR , Jr, Butter EM, Aman MG. Standardized Observation Analogue Procedure in the Treatment of Severe Childhood Aggression Study. J Child Adolesc Psychopharmacol. 2020 Feb;30(1):48-54. doi: 10.1089/cap.2019.0109. Epub 2019 Nov 15. PMID 31730370
- [Derived] Barterian JA, Arnold LE, Brown NV, Farmer CA, Williams C, Findling RL, Kolko DJ, Bukstein OG, Molina BSG, Townsend L, Aman MG. Clinical Implications From the Treatment of Severe Childhood Aggression (TOSCA) Study: A Re-Analysis and Integration of Findings. J Am Acad Child Adolesc Psychiatry. 2017 Dec;56(12):1026-1033. doi: 10.1016/j.jaac.2017.09.426. Epub 2017 Oct 6. PMID 29173736
- [Derived] Farmer CA, Epstein JN, Findling RL, Gadow KD, Arnold LE, Kipp H, Kolko DJ, Butter E, Schneider J, Bukstein OG, McNamara NK, Molina BS, Aman MG. Risperidone Added to Psychostimulant in Children with Severe Aggression and Attention-Deficit/Hyperactivity Disorder: Lack of Effect on Attention and Short-Term Memory. J Child Adolesc Psychopharmacol. 2017 Mar;27(2):117-124. doi: 10.1089/cap.2016.0040. Epub 2016 Jun 27. PMID 27348211
- [Derived] Gadow KD, Brown NV, Arnold LE, Buchan-Page KA, Bukstein OG, Butter E, Farmer CA, Findling RL, Kolko DJ, Molina BS, Rice RR Jr, Schneider J, Aman MG. Severely Aggressive Children Receiving Stimulant Medication Versus Stimulant and Risperidone: 12-Month Follow-Up of the TOSCA Trial. J Am Acad Child Adolesc Psychiatry. 2016 Jun;55(6):469-78. doi: 10.1016/j.jaac.2016.03.014. Epub 2016 Apr 13. PMID 27238065
- [Derived] Farmer CA, Arnold LE, Bukstein OG, Findling RL, Gadow KD, Li X, Butter EM, Aman MG. The treatment of severe child aggression (TOSCA) study: Design challenges. Child Adolesc Psychiatry Ment Health. 2011 Nov 10;5(1):36. doi: 10.1186/1753-2000-5-36. PMID 22074813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 256 participants were screened. 188 passed screening.
Pre-assignment Details: Between initial contact and randomization, 108 potential participants were lost for the following reasons: 68 subjects failed screen criteria, 4 were ineligible at Baseline, 10 withdrew consent, 4 were lost to follow-up, and 2 were unable to swallow medication.
Groups:
- Basic (Stimulant + PMT + Placebo): Children will receive active methylphenidate HCl and placebo. Parents will receive parent management training.
- Augmented (Stimulant + PMT + Risperidone): Children will receive active methylphenidate HCl and active risperidone. Parents will receive parent management training.
Period: Overall Study
Arm/Group | Basic (Stimulant + PMT + Placebo) | Augmented (Stimulant + PMT + Risperidone)
Started | 84 | 84
Completed | 71 | 66
Not Completed | 13 | 18

BASELINE CHARACTERISTICS:
Population: ADHD & severe physical aggression
Groups:
- Total: Total of all reporting groups
Arm/Group | Basic (Stimulant + PMT + Placebo) | Augmented (Stimulant + PMT + Risperidone) | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 84 | 84 | 168
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (1.98) | 9.0 (2.05) | 8.9 (2.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 64 | 65 | 129
Region of Enrollment [Number; unit: participants]
  United States | 84 | 84 | 168

OUTCOME MEASURES:

1. Primary Outcome: NCBRF-TIQ D-Total Score
Description: Parent ratings of aggression and hostility on the Nisonger Child Behavior Rating Form-Typical IQ (NCBRF-TIQ) D-Total Score. The NCBRF provides 1 prosocial subscale (Positive/Social) and 6 problem behavior subscales (Conduct Problem, Oppositional Behavior, Hyperactive, Inattentive, Overly Sensitive, and Withdrawn/Dysphoric). The NCBRF has excellent internal consistency, distinguishes between controls and subjects with DBDs. Conduct Problem and Oppositional Behavior subscales map closely to DSM-IV-TR symptoms of CD and ODD; they were scored together to form a variable called the D-Total.
  For the NCBRF D-Total, higher scores reflect worse behavior. Each subscale is scored by taking the rating (0 [did not occur or was not a problem] to 3 [occurred a lot or was a very severe problem]) for all component items. The D-Total score was computed by adding the 6 scores from the Oppositional subscale and the 10 items from the Conduct Problem subscale. Thus D-Total scores could range from 0-69.
Time Frame: Measured at baseline and Weeks 3, 4, 5, 6, 7, 8, 9
Population: ADHD & severe physical aggression
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Augmented (Stimulant + PMT + Risperidone): Children will receive active methylphenidate HCl and risperidone. Parents will receive parent management training
Arm/Group | Basic (Stimulant + PMT + Placebo) | Augmented (Stimulant + PMT + Risperidone)
Number analyzed (Participants) | 84 | 84
units on a scale
  Baseline | 43.5 (10.3) | 42.1 (10.4)
  Week 3 | 24.9 (15.3) | 25.9 (15.2)
  Week 4 | 22.4 (15.1) | 17.1 (12.5)
  Week 5 | 20.1 (15.7) | 12.1 (10.1)
  Week 6 | 20.7 (14.6) | 13.8 (12.1)
  Week 7 | 16.8 (12.8) | 13.0 (11.2)
  Week 8 | 17.8 (15.0) | 11.7 (10.2)
  Week 9 | 17.8 (15.4) | 10.7 (9.0)

2. Other Pre Specified Outcome: Antisocial Behavior Scale - Reactive Aggression Subscale
Description: The Antisocial Behavior Scale (ABS) is a 28-item scale that contains 10 Proactive Aggression items and six Reactive Aggression items. Each item is rated on a 3-point scale, ranging from 1 (Never) to 3 (Very often). Thus, scores on the Reactive Aggression subscale can range from 6 through 18; with higher scores indicating more reactive aggression.
Time Frame: Measured at baseline and Week 9
Population: ADHD & severe physical aggression
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Basic (Stimulant + PMT + Placebo) | Augmented (Stimulant + PMT + Risperidone)
Number analyzed (Participants) | 84 | 84
units on a scale
  Baseline | 15.9 (1.8) | 15.5 (2.4)
  Week 9 | 12.3 (3.1) | 11.0 (2.7)

3. Other Pre Specified Outcome: Clinical Global Impressions Scale for Improvement
Description: Using this clinician rating scale the patient's improvement is scored on a 7-point scale which ranges from "very much improved" (1), through "no change" (4), to "very much worse" (7). This scale was used at baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, & 9. Only endpoint (week 9 or subject's last visit) Clinical Global Impressions Scale for Improvement scores are reported below.
Time Frame: Measured at endpoint visit
Population: ADHD & severe physical aggression; participants who completed a study endpoint visit and were given a Clinical Global Impressions Scale for Improvement rating
Measure: Number; unit: participants
Arm/Group | Basic (Stimulant + PMT + Placebo) | Augmented (Stimulant + PMT + Risperidone)
Number analyzed (Participants) | 83 | 80
participants
  Much or very much improved at endpoint | 58 | 63
  Minimally improved at endpoint | 22 | 11
  Unchanged or worse at endpoint | 3 | 6

4. Other Pre Specified Outcome: Clinical Global Impressions Scale for Severity of Illness
Description: Using this clinician rating scale the severity of the illness is scored from 1= normal to 7= extremely ill. This scale was used at baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, & 9. Only endpoint (week 9 or subject's last visit) Clinical Global Impressions Scale for Severity of Illness scores are reported below.
Time Frame: Measured at endpoint visit
Population: ADHD and severe physical aggression; participants who completed a study endpoint visit and were given a Clinical Global Impressions Scale for Severity of Illness rating
Measure: Number; unit: participants
Arm/Group | Basic (Stimulant + PMT + Placebo) | Augmented (Stimulant + PMT + Risperidone)
Number analyzed (Participants) | 83 | 78
participants
  Normal/Borderline/Mildly ill at endpoint | 49 | 56
  Moderately/Markedly/Severely ill at endpoint | 34 | 22

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Only adverse events for weeks 4 to 9 (when the second medication was used) are reported. After subtracting the 22 participants who were not given the second medication, AE data were available for 80 basic treatment and 73 augmented treatment participants.
Arm/Group | Basic (Stimulant + PMT + Placebo) | Augmented (Stimulant + PMT + Risperidone)
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/73
Other Adverse Events (participants affected / at risk) | 69/80 | 62/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Basic (Stimulant + PMT + Placebo) (N=80) | Augmented (Stimulant + PMT + Risperidone) (N=73)
Trouble falling asleep (General disorders) | 29 | 14
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 14
Appetite decrease (Metabolism and nutrition disorders) | 19 | 9
Appetite increase (Metabolism and nutrition disorders) | 7 | 10
Diarrhea (Gastrointestinal disorders) | 9 | 5
Gastrointestinal discomfort (Gastrointestinal disorders) | 4 | 12
Vomiting (Gastrointestinal disorders) | 6 | 10
Sedation (General disorders) | 20 | 16
Headache (General disorders) | 17 | 16

LIMITATIONS AND CAVEATS:
These results were obtained with children selected for severity of aggression and disruptive behavior, and the risk-benefit ratio may well be decreased for children with milder disruptive behavior or no physical aggression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No